CLINICAL TRIAL: NCT03683550
Title: Randomized Trial Comparing Sentinel Lymph Node Excision (SLNE) With or Without Preoperative Hybrid Single-photon Emission Computed Tomography/Computed Tomography (SPECT/CT) in Melanoma
Brief Title: Comparing SLNE With or Without Preoperative Hybrid SPECT/CT in Melanoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Essen (Other)
Responsible Party: Principal Investigator, Dr. Joachim Klode, Prof. Dr. med, University Hospital, Essen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SNEPS 2018
Record Dates: First submitted 2018-09-20; First posted 2018-09-25 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Melanoma
Keywords: SLNE; SPECT/CT
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SPEC/CT (Experimental): SLNE with preoperative hybrid SPECT/CT
  Interventions: Procedure: SLNE with preoperative hybrid SPECT/CT
- Standard (Active Comparator): Standard SLNE (with planar preoperative lymphoscintigraphy)
  Interventions: Procedure: Standard SLNE

INTERVENTIONS:
Procedure: SLNE with preoperative hybrid SPECT/CT — Single-photon emission computed tomography/computed tomography (SPECT/CT) provides complementary functional and anatomical information and has been shown to be superior to planar imaging in a number of indications. It can provide valuable information before sentinel lymph node biopsy and advocate its use in a range of tumors such as truncal and head and neck melanomas.
  Arms: SPEC/CT
Procedure: Standard SLNE — The current gold standard for detection and targeted extirpation of the sentinel lymph node (SLN) is preoperative lymphoscintigraphy.
  Lymphoscintigraphy (sentinel lymph node mapping) is an imaging technique used to identify the lymph drainage basin, determine the number of sentinel nodes, differentiate sentinel nodes from subsequent nodes, locate the sentinel node in an unexpected location, and mark the sentinel node over the skin for biopsy.
  Arms: Standard

SUMMARY:
Melanoma has become a growing interdisciplinary problem in public health worldwide. It characteristically disseminates in an orderly progression through lymphatic channels to the regional lymph node and then to more distant sites.

Sentinel lymph node excision (SLNE) is probably the most important diagnostic and potentially therapeutic procedure for melanoma patients.

This is a randomized, open-label, multi-center, superiority, 2-parallel arms trial comparing sentinel lymph node excision with or without preoperative hybrid single photon emission computed tomography/computed tomography in patients with malignant melanoma.

DETAILED DESCRIPTION:
The presence of regional lymph node involvement is the single most important prognostic factor, lowering the 5-year survival rate to approximately 50%.

Recommendations for the use of SLNE for primary melanoma are included in the current American Joint Committee on Cancer guidelines. Critics argue that the routinely performed SLNE is a cost intensive surgical intervention with potential morbidity that does not offer patients any advantage in overall survival. The current gold standard for detection and targeted extirpation of the sentinel lymph node (SLN) is preoperative lymphoscintigraphy as an imaging technique to identify the lymph drainage basin, determine the number of sentinel nodes, differentiate sentinel nodes from subsequent nodes, locate the sentinel node in an unexpected location, and mark the sentinel node over the skin for biopsy. Single-photon emission computed tomography/computed tomography (SPECT/CT) provides complementary functional and anatomical information and has been shown to be superior to planar imaging in a number of indications. It can provide valuable information before sentinel lymph node biopsy and advocate its use in a range of tumors such as truncal and head and neck melanomas.

The objective of the planned multi-center randomized prospective trial is to compare distant metastasis-free survival (DMFS) in patients with cutaneous melanoma between sentinel lymph node excision with versus without preoperative SPECT/CT imaging and metastatic node detection.

ELIGIBILITY:
Inclusion Criteria:

* Patients with malignant melanoma in AJCC stages Ib / II
* Tumor depth of ≥1.0 mm
* Age ≥18 years to ≤75 years
* Have a primary melanoma that is cutaneous (including head, neck, trunk, extremity, scalp, palm, sole, subungual skin tissues
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* Life expectancy of at least 5 years from the time of diagnosis, not considering the melanoma in question, as determined by the principal investigator (PI)
* Willing to return to the trial center for follow-up examinations and procedures as outlined in the protocol
* Randomization must be completed no more than 120 days following the diagnostic biopsy of the primary melanoma
* Negative pregnancy test for female and effective contraception for both male and female subjects if the risk of conception exists
* Signed written informed consent prior to the performance of any trial specific procedure

Exclusion Criteria:

* History of previous or concurrent (i.e., second primary) invasive melanoma
* Primary melanoma of the eye, mucous membranes or internal viscera
* Any additional solid tumor or hematologic malignancy during the past 5 years except skin lesions of squamous cell carcinoma, basal cell carcinoma, or uterine cervical cancer
* Skin grafts, tissue transfers or flaps that have the potential to alter the lymphatic drainage pattern from the primary melanoma to a lymph node basin
* Hypersensitivity to the active substance(s), to any of the excipients or to any of the components of the labelled radiopharmaceutical
* Extensive previous surgery in the region of the primary tumor site or complete lymph node dissection (CLNDs) or sentinel lymphadenectomy (SLs) (before evaluation of the current melanoma) that may have altered the lymphatic drainage pattern from the primary cutaneous melanoma to a potential lymph node basin
* Organic brain syndrome or significant impairment of basal cognitive function or any psychiatric disorder that might preclude participation in the full protocol, or be exacerbated by therapy (e.g., severe depression)
* Pregnancy (absence to be confirmed by ß-human chorionic gonadotropin test) or lactation period
* Medical or psychological conditions that would not permit the subject to complete the study or sign informed consent
* Known alcohol or drug abuse
* Participation in another clinical study within the 30 days before registration
* Significant disease which, in the investigator's opinion, would exclude the patient from the study
* Legal incapacity or limited legal capacity

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 836 (Estimated)
Dates: Start 2018-09-25 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Distant free metastasis survival (DFMS) | 6 years
  The number of patients free of distant metastasis after randomization in arm A compared to DFMS in arm B.

SECONDARY OUTCOMES:
Overall survival (OS) | 6 years
  Overall Survival (OS) of a patient defined as the time frame start of run-in phase until documented date of death
Disease-free survival (DFS) | 6 years
  The number of patients alive and free of disease after randomization in arm A compared to DFS in arm B.
False negative rate of SLN | 3 years
  Rate of local relapse within a 12 month follow-up period (false negative rate of sentinel lymph nodes [SLN])
Sensitivity | 3 years
  Number of positive SLN
Complication rate | 6 years
  Intraoperative and postoperative complications due to SLNE
Quality of Life (QoL) | 6 years
  Measure of health outcome by questionnaire. The EuroQol-5 Dimensions-5 Level (EQ-5D-5L) questionnaire consists of five HrQoL dimensions (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression), with each dimension specifying five levels of severity [no (level 1), slight (level 2), moderate (level 3), severe (level 4), and extreme problems/unable (level 5)], which allows the description of 3125 health states.
Quality adjusted life years (QALY) | 6 years
  Assessing the health economic relevance
Number of inpatient days | 6 years
  To calculate the cost of the two treatment options the number of inpatient days will be counted and compared for each treatment arm.
Overall costs during hospital stays | 6 years
  Overall costs during hospital stays will be summed up and compared.
Incidence of Treatment-Emergent Adverse Events | 6 years
  Intervention-related safety events will be documented during the trial period

CONTACTS AND LOCATIONS:
Overall Officials: Ingo Stoffels, MD, Principal Investigator — Department of Dermatology, University Hospital Essen; Joachim Klode, MD, Principal Investigator — Department of Dermatology, University Hospital Essen
Locations (13):
- Germany (13):
  - Department of Dermatology, University Hospital Essen, Essen, North Rhine-Westphalia
  - Hospital Augsburg, Department of Dermatology, Augsburg
  - Vivantes Hospital Berlin Neukölln, Berlin
  - University Hospital Bonn, Bonn
  - Hospital Dresden Friedrichstadt, Department of Dermatology and Allergology, Dresden
  - Universitätsklinik Dresden, Dresden
  - Universitätskliniken Düsseldorf, Düsseldorf
  - Universitätsklinikum Giessen, Giessen
  - University Hospital Göttingen, Department of Dermatology, Göttingen
  - Universitätsklinikum Hamburg Eppendorf, Hamburg
  - University Hospital Heidelberg, Department of Dermatology, Heidelberg
  - University Hospital Lübeck, Department of Dermatology, Lübeck
  - University Hospital Tübingen, Tübingen

REFERENCES:
- [Derived] Stoffels I, Herrmann K, Rekowski J, Jansen P, Schadendorf D, Stang A, Klode J. Sentinel lymph node excision with or without preoperative hybrid single-photon emission computed tomography/computed tomography (SPECT/CT) in melanoma: study protocol for a multicentric randomized controlled trial. Trials. 2019 Feb 4;20(1):99. doi: 10.1186/s13063-019-3197-7. PMID 30717811